CLINICAL TRIAL: NCT01667614
Title: Comparison of Efficacy of Losartan/Spironolactone and Losartan/Enalapril on Urinary Albumin Excretion, Estimated Glomerular Filtration Rate, and Blood Pressure in Patients With Type 2 Diabetes Nephropathy
Brief Title: Effects of Spironolactone Combination Therapy on Proteinuria, Kidney Function, and Blood Pressure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Alireza Esteghamati, Professor Alireza Esteghamati, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 90-2-27-16-10
Record Dates: First submitted 2012-08-15; First posted 2012-08-17 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2012-08

CONDITIONS: Type 2 Diabetes Mellitus; Diabetic Nephropathy; Essential Hypertension
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Nephropathies; Essential Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACE/ARB (No Intervention): In 62 patients previously treated with enalapril (10-30 mg daily) + losartan (50-100 mg daily), this regimen was continued.
- Spironolactone/ARB (Active Comparator): spironolacone 25 mg tablets added to losartan
  Interventions: Drug: spironolacone 25 mg tablets added to losartan

INTERVENTIONS:
Drug: spironolacone 25 mg tablets added to losartan — spironolactone 25 mg once daily added to losartan
  Arms: Spironolactone/ARB

SUMMARY:
The detrimental effects of aldostrone are not adequately arrested by the use of angiotensin converting enzyme (ACE), angiotensin II receptor blocker (ARB) or a combination of both. Recent evidence has provided robust evidence that aldostrone escape plays an important role in this regard. It is believed that aldostrone escape occurs quite commonly with reports indicating prevalence rates as high as 22% with ARBs and 40% with ACE inhibitors. In a trial of patients with diabetes and hypertension it was shown that treatment of aldostrone escape with spironolactone 25 mg daily for three months significantly reduces proteinuria. A number of other trials have similarly observed that addition of spironolactone to an ACE inhibitor based regimen provides additional benefits on proteinuria reduction, blood pressure control, and prevention of glomerular filtration rate (GFR) decline. Most of the available trials in this regard are of short duration (e.g. three months), and have added spironolactone to an ACE or ACE+ARB based regimen (the so-called triple blockade). Currently, evidence evaluating efficacy of a combined ARB+spironolactone regimen compared with conventional double RAS blockade (i.e. ACE+ARB) is lacking. Hence, this randomized open label trial was initiated to determine the effects of addition of spironolactone 25 mg daily to losartan over a period of 18 months.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes patients with diabetic nephropathy in the range of micro- or macroalbuminuria
* treatment with combination of enalapril and losartan for more than one year

Exclusion Criteria:

* history of non-adherence to prescribed medication assessed by the prescribing physician
* baseline potassium > 5.5 meq/L
* chronic kidney disease stages 4 or 5
* history or evidence of non-diabetic kidney disease

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2010-05; Primary Completion 2012-03 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Urinary albumin excretion | 18 months
  Urinary albumin excretion assessed by overnight (12 hour) collection of urine. Measured at baseline, 3rd month, 6th month, 9th month, 12th month, 15th month, and 18th month.

SECONDARY OUTCOMES:
estimated glomerular filtration rate | 18 months
  estimated glomerular filtration rate calculated using the formula developed by Chronic Kidney Disease Epidemiology Collaboration. Measured at baseline, 3rd month, 6th month, 9th month, 12th month, 15th month, and 18th month.
Blood pressure | 18 months
  Systolic and diastolic blood pressure assessed by mercury sphygnomanometry. Patients were placed in a sitting position and after ten minutes rest, two readings from right-side hand with five minutes interval were obtained. Measured at baseline, 3rd month, 6th month, 9th month, 12th month, 15th month, and 18th month.
serum creatinine concentrations | 18 months
  serum creatinine concentrations assessed by Jaffe method. Measured at baseline, 3rd month, 6th month, 9th month, 12th month, 15th month, and 18th month.
Serum potassium concentrations | 18 months
  Serum potassium concentrations measured at baseline, 1st month, 3rd month, 6th month, 9th month, 12th month, 15th month, and 18th month.

CONTACTS AND LOCATIONS:
Overall Officials: Alireza Esteghamati, M.D., Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Tehran University of Medical Sciences, Vali-asr hospital, Endocrinology and Metabolism Research Center, Tehran, Tehran Province, Iran

REFERENCES:
- [Derived] Chung EY, Ruospo M, Natale P, Bolignano D, Navaneethan SD, Palmer SC, Strippoli GF. Aldosterone antagonists in addition to renin angiotensin system antagonists for preventing the progression of chronic kidney disease. Cochrane Database Syst Rev. 2020 Oct 27;10(10):CD007004. doi: 10.1002/14651858.CD007004.pub4. PMID 33107592